CLINICAL TRIAL: NCT02389439
Title: Monitoring and Evaluation of the Therapeutic Efficacy and Safety of Pyronaridine-artesunate for the Treatment of Uncomplicated Falciparum Malaria in Western Cambodia, an Area of Artemisinin-resistant Falciparum Malaria
Brief Title: Efficacy and Safety of Pyronaridine-artesunate for the Treatment in Uncomplicated Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: NCHADS - Ministry of Health of Cambodia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cambodia1
Record Dates: First submitted 2015-01-29; First posted 2015-03-17 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2015-04

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyronaridine-artesunate (Experimental): Pyronaridine-artesunate (Pyramax®, Shin Poong Pharmaceuticals). One tablet contains 60mg artesunate+ 180mg pyronaridine. Dosing will be according to body weight.
  It will be taken orally with water, once daily for 3 days. Each dose will be administered under the supervision. A dose will be repeated in full if vomiting occurs within 30 minutes of administration of the first day of administration only.
  20 - < 24 kg = 1 tab 24 - < 45 kg = 2 tabs 45 - < 65 kg = 3 tabs 65 and above = 4 tabs
  Interventions: Drug: Pyronaridine-artesunate

INTERVENTIONS:
Drug: Pyronaridine-artesunate
  Other Names: Pyramax

SUMMARY:
This study is a prospective, single arm, open-labelled clinical trial. The total number subjects will be 145 patients to receive Pyronaridine-artesunate once daily for 3 days. Dosing will be according to the body weight.

All patients will have a blood smear examined daily during the first week by microscopy until parasite clearance (2 consecutive negative slides on two consecutive days; both asexual and sexual stages). A negative blood slide will be defined as parasite count negative per 1000 WBC in two consecutive days. The sample on day 3 will be taken as close as possible to 72h after the initial blood smear.

Participant will follow up for 42 days to assess the drug efficacy and safety (Day 7, 14, 21, 28, 35 and 42).

ELIGIBILITY:
Inclusion Criteria:

* Adults and children ≥ 20 kg
* Symptomatic of malaria infection, i.e. history of fever within 24 hours and/or presence of fever >37.5°c.
* Microscopic confirmation of asexual stages of P. falciparum (P. falciparum and mixed infection in Pailin only)
* Capability of taking an oral medication
* Written informed consent given to participate in the trial
* Willingness and ability to adhere to follow-up visit schedule

Exclusion Criteria:

* Pregnancy or lactation (urine test for β HCG to be performed on any woman of child bearing age, that is 18 to 45 y/o)
* Female aged 12-18y
* Parasitemia > 150 000/µL).
* Signs or symptoms indicative of severe malaria:

  * Impaired consciousness (Blantyre Coma Score <5)
  * Severe anaemia (Hct<15%)
  * Bleeding disorder -evidenced by epistaxis, bleeding gums, frank haematuria, bleeding from venepuncture sites
  * Respiratory distress
  * Severe jaundice
* Known hypersensitivity to artemisinins - defined as history of erythroderma/other severe cutaneous reaction, angioedema or to pyronaridine
* History of splenectomy
* Known history or evidence of clinically significant disorders, such as:

  * Known active Hepatitis A, e.g. by detection of anti HAV-IgM.
  * Known hepatitis B surface antigen (HBsAg) carrier.
  * Known hepatitis C antibody (HCV Ab).
  * Liver function tests (AST/ALT levels) more than 2.5 times the upper limit of normal range.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
result of PCR | 42 day

SECONDARY OUTCOMES:
hepatic biological values | at day 0, 3,7 and day 28
  the hepatic biological values will be measured which are AST,ALT,albumin and total bilirubin
eosinophil count | at day 0, 3, 7 and day 28
K13 and pfmdr1 of P falciparum resistance | at day 0, 3, 7 and day 28
numbers of patients with a positive malaria slide 72 hours after treatment initiation | 72 hours
fever clearance time | 24 hours
  the time taken for tympanic temperature to fall below 37.5˚C and remain there for at least 24 hours
Number of patient with reinfection and recrudescences | over 42 days
PCR uncorrected ACPR | at 28 days or 42 days
  PCR uncorrected ACPR at 28 days or 42 days for P. falciparum, P. falciparum and mixed infections in Pailin
PCR corrected ACPR | at 28 days and 42 days
  PCR corrected ACPR at 28 days or for P. falciparum, P. vivax and mixed infections and at 42 days for P. falciparum and mixed infections
Gametocyte carriage rates | at day 0, 3, 7 day 28
gametocyte clearance times | at day 0, 3, 7 and day28

CONTACTS AND LOCATIONS:
Locations (3):
- Cambodia (3):
  - Tasanh Health Centre, Battambang, Battambang
  - Referral hospital (Pailin), Pailin
  - Promoy Health Centre (Pursat), Pursat

REFERENCES:
- [Derived] Leang R, Canavati SE, Khim N, Vestergaard LS, Borghini Fuhrer I, Kim S, Denis MB, Heng P, Tol B, Huy R, Duparc S, Dondorp AM, Menard D, Ringwald P. Efficacy and Safety of Pyronaridine-Artesunate for Treatment of Uncomplicated Plasmodium falciparum Malaria in Western Cambodia. Antimicrob Agents Chemother. 2016 Jun 20;60(7):3884-90. doi: 10.1128/AAC.00039-16. Print 2016 Jul. PMID 26926629